CLINICAL TRIAL: NCT03131687
Title: A Phase 2 Study of Once-Weekly LY3298176 Compared With Placebo and Dulaglutide in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16335; I8F-MC-GPGB (Other: Eli Lilly and Company); 2016-004179-33 (EudraCT Number)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Tirzepatide placebo and dulaglutide placebo administered subcutaneously (SC) once weekly.
  Interventions: Drug: Placebo
- 1 mg Tirzepatide (Experimental): 1 milligrams (mg) tirzepatide administered SC once weekly. Dulaglutide placebo administered SC once weekly.
  Interventions: Drug: tirzepatide; Drug: Placebo
- 5 mg Tirzepatide (Experimental): 5 mg tirzepatide administered SC once weekly. Dulaglutide placebo administered SC once weekly.
  Interventions: Drug: tirzepatide; Drug: Placebo
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once weekly. Dulaglutide placebo administered SC once weekly.
  Interventions: Drug: tirzepatide; Drug: Placebo
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once weekly. Dulaglutide placebo administered SC once weekly.
  Interventions: Drug: tirzepatide; Drug: Placebo
- 1.5 mg Dulaglutide (Active Comparator): 1.5 mg Dulaglutide administered SC once weekly. Tirzepatide placebo administered SC once weekly.
  Interventions: Drug: Dulaglutide; Drug: Placebo

INTERVENTIONS:
Drug: tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 1 mg Tirzepatide; 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 1.5 mg Dulaglutide
Drug: Placebo — Administered SC

SUMMARY:
The purpose of this study is to evaluate the efficacy of the study drug tirzepatide in participants with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Have had type 2 diabetes (T2D) for ≥6 months according to the World Health Organization (WHO) classification.
* Have HbA1c of 7.0% to 10.5%, inclusive, as assessed by the central laboratory.
* If on metformin, have been treated with stable doses of metformin for at least 3 months.
* Have a body mass index (BMI) ≥23 and <50 kilograms per square meter.

Exclusion Criteria:

* Have type 1 diabetes (T1D).
* Have used any glucose-lowering medication other than metformin within 3 months prior to study entry or during screening/lead-in period or have used any glucagon-like peptide-1 receptor agonists (GLP-1 RAs) at any time in the past.
* Have had any of the following cardiovascular conditions: acute myocardial infarction (MI), New York Heart Association Class III or Class IV heart failure, or cerebrovascular accident (stroke).
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine aminotransferase (ALT) level >2.5 times the upper limit of the reference range, as determined by the central laboratory at study entry; participants with NAFLD are eligible for participation in this trial.
* Have had chronic or acute pancreatitis any time prior to study entry.
* Have an estimated glomerular filtration rate (eGFR) <45 milliliters/minute/1.73 square meter, calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation.
* Have serum calcitonin ≥20 picograms per milliliter, as determined by the central laboratory at study entry.
* Have any condition that is a contraindication for use of the GLP-1 RA class (per country-specific labels) at study entry or develop such condition between study entry and randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (35):
  - Internal Medicine Center LLC, Mobile, Alabama
  - Anaheim Clinical Trails, Anaheim, California
  - Valley Research, Fresno, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Valley Clinical Trails, Inc, Northridge, California
  - Artemis Institute For Clinical Research, San Diego, California
  - Artemis Institute For Clinical Research, San Marcos, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators INC, Tustin, California
  - Chase Medical Research, Waterbury, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - East Coast Institute For Research, Jacksonville, Florida
  - Suncoast Research Group, LCC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Palm Harbor Medical Associate, Palm Harbor, Florida
  - Solaris Clinical Research, Meridian, Idaho
  - Iderc P.L.C., West Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrine, Topeka, Kansas
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Clinical Research Professionals, St Louis, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Premier Research, Trenton, New Jersey
  - Manhattan Medical Research, New York, New York
  - Lillestol Research LLC, Fargo, North Dakota
  - Aventiv Research, Columbus, Ohio
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - PMG Research Of Charleston LLC, Moncks Corner, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - PMG Research Of Knoxville, Knoxville, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Chrysalis Clinical Research, St. George, Utah
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Gdansk
  - "For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician.", Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Katowice
  - Clinica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária LTDA, Lodz
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Szczecin
- Puerto Rico (3):
  - Manati Center for Clinical Research, Manatí, PR
  - Clinical Research Puerto Rico. Inc, San Juan
  - GCM Medical Group PSC, San Juan
- Slovakia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malacky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Púchov
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Trenčín
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Trenčín

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595
- [Derived] Pirro V, Roth KD, Lin Y, Willency JA, Milligan PL, Wilson JM, Ruotolo G, Haupt A, Newgard CB, Duffin KL. Effects of Tirzepatide, a Dual GIP and GLP-1 RA, on Lipid and Metabolite Profiles in Subjects With Type 2 Diabetes. J Clin Endocrinol Metab. 2022 Jan 18;107(2):363-378. doi: 10.1210/clinem/dgab722. PMID 34608929
- [Derived] Hartman ML, Sanyal AJ, Loomba R, Wilson JM, Nikooienejad A, Bray R, Karanikas CA, Duffin KL, Robins DA, Haupt A. Effects of Novel Dual GIP and GLP-1 Receptor Agonist Tirzepatide on Biomarkers of Nonalcoholic Steatohepatitis in Patients With Type 2 Diabetes. Diabetes Care. 2020 Jun;43(6):1352-1355. doi: 10.2337/dc19-1892. Epub 2020 Apr 14. PMID 32291277
- [Derived] Frias JP, Nauck MA, Van J, Kutner ME, Cui X, Benson C, Urva S, Gimeno RE, Milicevic Z, Robins D, Haupt A. Efficacy and safety of LY3298176, a novel dual GIP and GLP-1 receptor agonist, in patients with type 2 diabetes: a randomised, placebo-controlled and active comparator-controlled phase 2 trial. Lancet. 2018 Nov 17;392(10160):2180-2193. doi: 10.1016/S0140-6736(18)32260-8. Epub 2018 Oct 4. PMID 30293770
- See also: A Study of tirzepatide in Participants With Type 2 Diabetes Mellitus — https://www.lillytrialguide.com/en-US/studies/diabetes/GPGB#?postal=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Started | 51 | 53 | 55 | 52 | 53 | 54
Received at Least One Dose of Study Drug | 51 | 52 | 55 | 51 | 53 | 54
Completed | 45 | 44 | 52 | 48 | 45 | 49
Not Completed | 6 | 9 | 3 | 4 | 8 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 2 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 4 | 0 | 1 | 4 | 2
Not completed — Participant Started New Diabetic Drug | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Principle Investigator Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Inadvertent Enrollment | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 1 mg Tirzepatide: 1 mg tirzepatide administered SC once weekly. Dulaglutide placebo administered SC once weekly.
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide | Total
Number analyzed (Participants) | 51 | 52 | 55 | 51 | 53 | 54 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (8.85) | 57.4 (8.85) | 57.9 (8.22) | 56.5 (9.92) | 56.0 (7.58) | 58.7 (7.81) | 57.2 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 21 | 21 | 31 | 30 | 148
  Male | 29 | 29 | 34 | 30 | 22 | 24 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 25 | 22 | 26 | 23 | 19 | 142
  Not Hispanic or Latino | 19 | 23 | 23 | 20 | 27 | 27 | 139
  Unknown or Not Reported | 5 | 4 | 10 | 5 | 3 | 8 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 1 | 2 | 2 | 1 | 15
  Asian | 1 | 0 | 0 | 1 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Black or African American | 2 | 5 | 6 | 7 | 6 | 4 | 30
  White | 41 | 42 | 46 | 37 | 43 | 44 | 253
  More than one race | 2 | 1 | 2 | 2 | 0 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 4 | 4 | 3 | 3 | 1 | 1 | 16
  United States | 36 | 37 | 38 | 37 | 43 | 43 | 234
  Poland | 6 | 7 | 4 | 6 | 6 | 2 | 31
  Slovakia | 5 | 4 | 10 | 5 | 3 | 8 | 35
Hemoglobin A1C (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.04 (0.861) | 8.21 (0.905) | 8.17 (0.961) | 8.15 (1.072) | 8.13 (1.061) | 8.13 (0.954) | 8.14 (0.966)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Hemoglobin A1c (HbA1c) Bayesian Dose Response
Description: HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.This was a Bayesian dose response analysis of HbA1c (%) change from baseline. At baseline: Mean (SD = Standard Deviation) of baseline HbA1c (%). After baseline: Posterior Mean (SD = Posterior Standard Deviation) of HbA1c (%) change from baseline.
  The Least Squares Mean is Posterior mean.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline excluding data after rescue drug initiation.
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 44 | 45 | 52 | 47 | 44 | 49
Percentage of HbA1c | -0.06 (0.14) | -1.06 (0.11) | -1.73 (0.08) | -1.89 (0.08) | -1.94 (0.09) | -1.21 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.00, Standard Deviation 0.17 — Statistics are estimated from a Bayesian hierarchical logistic dose response model along with a titrated integrated two-component prediction model to estimate missing values
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.67, Standard Deviation 0.17 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.83, Standard Deviation 0.17 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.89, Standard Deviation 0.17 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline to Week 12 in Hemoglobin A1c (HbA1c) Bayesian Dose Response
Description: HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. This was a Bayesian dose response analysis of HbA1c (%) change from baseline. At baseline: Mean (SD = Standard Deviation) of baseline HbA1c (%). After baseline: Posterior Mean (SD = Posterior Standard Deviation) of HbA1c (%) change from baseline.
  The Least Squares Mean is Posterior mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value excluding data after rescue drug initiation.
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 48 | 45 | 52 | 48 | 48 | 51
Percentage of HbA1c | -0.05 (0.13) | -0.94 (0.10) | -1.54 (0.07) | -1.68 (0.08) | -1.72 (0.08) | -1.08 (0.13)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -0.89, Standard Deviation 0.15 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.49, Standard Deviation 0.15 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.62, Standard Deviation 0.15 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; Posterior Mean Difference = -1.67, Standard Deviation 0.15 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline to Week 26 in HbA1c
Description: HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. The Least Squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included the independent variables: Baseline + Baseline BMI Group + Baseline Metformin Flag + Treatment + Time + Treatment*Time.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug who had a baseline and postbaseline value excluding data after study drug discontinuation or rescue drug initiation.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 41 | 44 | 47 | 43 | 35 | 47
Percentage of HbA1c | 0.1 (0.16) | -0.7 (0.16) | -1.6 (0.15) | -2.0 (0.16) | -2.4 (0.17) | -1.1 (0.15)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.4]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -1.7, 95% CI 2-sided [-2.2 to -1.3]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -2.1, 95% CI 2-sided [-2.5 to -1.6]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -2.5, 95% CI 2-sided [-2.9 to -2.0]

4. Secondary Outcome: Change From Baseline to Week 12 in HbA1c
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: randomized participants who received at least one dose of study drug who had a baseline and postbaseline value excluding data after study drug discontinuation or rescue drug initiation.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 44 | 44 | 49 | 47 | 36 | 49
Percentage of HbA1c | -0.1 (0.13) | -0.9 (0.13) | -1.7 (0.13) | -2.0 (0.13) | -2.1 (0.15) | -1.2 (0.13)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.4]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.0 to -1.3]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.3 to -1.5]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-2.4 to -1.7]

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with independent variables: Baseline + Baseline HbA1C Group + Baseline BMI Group + Baseline Metformin Flag + Treatment + Time + Treatment*Time.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value excluding data after study drug discontinuation or rescue drug initiation.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (Kg)
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 41 | 44 | 48 | 44 | 35 | 47
Kilograms (Kg) | -0.4 (0.81) | -0.9 (0.80) | -4.8 (0.77) | -8.7 (0.80) | -11.3 (0.88) | -2.7 (0.78)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.655, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.7 to 1.7]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-6.6 to -2.3]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-10.5 to -6.0]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -10.9, 95% CI 2-sided [-13.3 to -8.6]

6. Secondary Outcome: Percentage of Participants With 5% or Greater Body Weight Loss From Baseline
Description: Percentage of participants with 5% or greater body weight loss from baseline last observation carried forward (LOCF) analyses using Logistic regression model with Baseline value + Baseline HbA1C Group + Baseline BMI Group + Baseline Metformin + Treatment as factors.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52 | 55 | 51 | 53 | 54
percentage of participants | 0 | 13.5 | 47.3 | 70.6 | 62.3 | 22.2
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.053, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p = 0.002, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic

7. Secondary Outcome: Percentage of Participants With 10% or Greater Body Weight Loss From Baseline
Description: Percentage of participants with 10% or greater body weight loss from baseline LOCF analyses using Logistic regression model with Baseline value + Baseline HbA1C Group + Baseline BMI Group + Baseline Metformin + Treatment as factors.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52 | 55 | 51 | 53 | 54
percentage of participants | 0 | 5.8 | 16.4 | 39.2 | 37.7 | 9.3
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.193, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p = 0.036, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p = 0.003, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p = 0.003, Regression, Logistic

8. Secondary Outcome: Percentage of Participants Reaching the HbA1c Target of ≤6.5%
Description: Percentage of participants with HbA1c ≤6.5% at Week 26 using a logistic regression model for endpoint used last observation carried forward (LOCF) method including baseline value, baseline BMI Group, baseline Metformin and treatment as factors.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug excluding data after study drug discontinuation or rescue drug initiation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52 | 55 | 50 | 53 | 54
percentage of participants | 2.0 | 15.4 | 63.6 | 82.0 | 58.5 | 38.9
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.030, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic

9. Secondary Outcome: Percentage of Participants Reaching the HbA1c Target of <7.0%
Description: Percentage of participants with HbA1c <7.0% at Week 26 using a logistic regression model for endpoint used last observation carried forward (LOCF) method including baseline value, baseline BMI Group, baseline Metformin and treatment as factors.
Time Frame: Week 26
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Groups:
- 1 mg Tirzepatide: 1 mg tirzepatide administered SC. Dulaglutide placebo administered SC once weekly.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52 | 55 | 50 | 53 | 54
percentage of participants | 11.8 | 32.7 | 69.1 | 90.0 | 77.4 | 51.9
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.008, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Regression, Logistic

10. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates: Baseline + Baseline HbA1C Group + Baseline BMI Group + Baseline Metformin Flag + Treatment + Time + Treatment*Time.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Groups:
- 5 mg Tirzepatide: 5 mg tirzepatide administered SC. Dulaglutide placebo administered SC.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 40 | 44 | 48 | 44 | 35 | 46
milligrams per deciliter (mg/dL) | 15.5 (6.66) | -6.8 (6.43) | -40.7 (6.23) | -60.7 (6.36) | -57.5 (7.10) | -21.2 (6.40)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -22.4, 95% CI 2-sided [-39.4 to -5.3]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -56.2, 95% CI 2-sided [-72.9 to -39.5]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = -76.3, 95% CI 2-sided [-93.3 to -59.2]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -73.0, 95% CI 2-sided [-90.9 to -55.2]

11. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C)
Description: LS means were calculated using MMRM model with independent variables: Baseline, Baseline HbA1C Group, Baseline BMI Group, Baseline Metformin Flag,Treatment, time, treatment*time.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value.
Measure: Least Squares Mean (Standard Error); unit: Millimoles Per Litre (mmol/L)
Groups:
- 5 mg Tirzepatide: 5 mg tirzepatide administered SC. Dulaglutide placebo administered SC once weekly.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 45 | 46 | 53 | 48 | 46 | 51
Millimoles Per Litre (mmol/L) | 0.0 (0.03) | -0.0 (0.03) | 0.0 (0.03) | 0.0 (0.03) | 0.1 (0.03) | 0.0 (0.03)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.396, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p = 0.903, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p = 0.536, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p = 0.325, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.1]

12. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: LS means were calculated using MMRM model with independent variables: Baseline, Baseline HbA1C Group, Baseline BMI Group, Baseline Metformin Flag, Treatment, Time, Treatment*Time.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value.
Measure: Least Squares Mean (Standard Error); unit: Millimoles Per Litre (mmol/L)
Groups:
- 1.5 mg Dulaglutide: 1.5 mg Dulaglutide administered SC. Tirzepatide placebo administered SC.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 45 | 46 | 53 | 48 | 46 | 51
Millimoles Per Litre (mmol/L) | 0.3 (0.13) | 0.2 (0.13) | -0.1 (0.12) | -0.3 (0.12) | -0.3 (0.13) | -0.2 (0.12)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.565, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.1]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p = 0.001, Mixed Models Analysis; Median Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.3]

13. Secondary Outcome: Change From Baseline in Triglycerides
Description: as for outcome 12
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value.
Measure: Least Squares Mean (Standard Error); unit: Millimoles Per Litre (mmol/L)
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 45 | 46 | 53 | 48 | 46 | 51
Millimoles Per Litre (mmol/L) | 0.3 (0.16) | -0.0 (0.16) | -0.5 (0.15) | -0.7 (0.15) | -0.8 (0.16) | -0.3 (0.15)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.164, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.4]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.4 to -0.6]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -1.1, 95% CI 2-sided [-1.5 to -0.7]

14. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C)
Description: as for outcome 12
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value.
Measure: Least Squares Mean (Standard Error); unit: Millimoles Per Litre (mmol/L)
Groups:
- Placebo: Tirzepatide placebo and dulaglutide placebo administered SC once weekly.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 42 | 45 | 52 | 48 | 45 | 50
Millimoles Per Litre (mmol/L) | 0.2 (0.12) | 0.2 (0.11) | 0.0 (0.11) | -0.0 (0.11) | -0.1 (0.12) | -0.1 (0.11)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.919, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p = 0.194, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p = 0.145, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p = 0.067, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.0]

15. Secondary Outcome: Change From Baseline in Waist Circumference
Description: as for outcome 12
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had a baseline and postbaseline value.
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 42 | 44 | 47 | 44 | 35 | 47
centimeters (cm) | -1.3 (0.91) | -2.1 (0.89) | -5.1 (0.86) | -7.4 (0.88) | -10.2 (1.00) | -2.5 (0.87)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Tirzepatide; Test type: Other; p = 0.539, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.1 to 1.6]
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tirzepatide; Test type: Other; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-6.1 to -1.5]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-8.4 to -3.7]
Statistical Analysis 4: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-11.3 to -6.4]

16. Secondary Outcome: Number of Participants With Anti-Drug Antibodies
Description: Number of Participants With Anti-Drug Antibodies.
Time Frame: Baseline through Week 30
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Tirzepatide placebo and dulaglutide placebo administered subcutaneously (SC).
- 1 mg Tirzepatide: 1 mg tirzepatide administered SC. Dulaglutide placebo administered SC.
- 10 mg Tirzepatide: 10 mg tirzepatide administered SC. Dulaglutide placebo administered SC.
- 15 mg Tirzepatide: 15 mg tirzepatide administered SC. Dulaglutide placebo administered SC.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52 | 55 | 51 | 53 | 54
Participants | 0 | 16 | 19 | 24 | 26 | 0

17. Secondary Outcome: Pharmacokinetics (PK): Model Predicted Concentration at Steady State (Css) of Tirzepatide
Description: Pharmacokinetics (PK): Model Predicted Concentration at Steady State (Css) of Tirzepatide
Time Frame: Predose: Week 1,8,12 and 26; Postdose: Week 1,2,4 and 12
Population: All randomized participants who received at least one dose of Tirzepatide study drug excluding post rescue data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms Per Millilitre (ng/mL)
Arm/Group | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 52 | 55 | 51 | 53
Nanograms Per Millilitre (ng/mL) | 78.6 (29) | 394 (29) | 787 (29) | 1180 (29)

ADVERSE EVENTS:
Time Frame: Up To 34 Weeks
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Tirzepatide placebo and dulaglutide placebo administered (SC) once weekly.
- 1 mg Tirzepatide: 1 mg tirzepatide and placebo given SC once weekly.
- 15 mg Tirzepatide + Placebo: 15 mg tirzepatide administered SC once weekly. Dulaglutide placebo administered SC once weekly.
Arm/Group | Placebo | 1 mg Tirzepatide | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide + Placebo | 1.5 mg Dulaglutide
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/52 | 0/55 | 0/51 | 0/53 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/51 | 2/52 | 1/55 | 3/51 | 2/53 | 3/54
Other Adverse Events (participants affected / at risk) | 17/51 | 17/52 | 29/55 | 32/51 | 39/53 | 31/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | 1 mg Tirzepatide (N=52) | 5 mg Tirzepatide (N=55) | 10 mg Tirzepatide (N=51) | 15 mg Tirzepatide + Placebo (N=53) | 1.5 mg Dulaglutide (N=54)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | 1 mg Tirzepatide (N=52) | 5 mg Tirzepatide (N=55) | 10 mg Tirzepatide (N=51) | 15 mg Tirzepatide + Placebo (N=53) | 1.5 mg Dulaglutide (N=54)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 4 (7) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 4 (4) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (13) | 13 (17) | 12 (13) | 17 (23) | 9 (12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 6 (7) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 11 (17) | 11 (13) | 21 (29) | 16 (22)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (8) | 8 (9) | 14 (20) | 5 (6)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (2) | 3 (3) | 2 (5) | 3 (6) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 2 (3) | 1 (1) | 4 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 4 (7) | 1 (3) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 4 (7) | 2 (3) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 11 (12) | 13 (14) | 10 (13) | 3 (3)
Dizziness (Nervous system disorders) | 2 (3) | 4 (4) | 2 (2) | 2 (2) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT03131687/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT03131687/SAP_001.pdf